CLINICAL TRIAL: NCT00636090
Title: Molecular, Genetic, and Genomic Assessments of MTOR Inhibition in Metastatic Hormone-Refractory Prostate Cancer Tissue From Patients Treated With RAD001
Brief Title: Molecular, Genetic, and Genomic Assessments From Patients Treated With RAD001
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: Pro00000346; CA123175; R01-A2-022207
Record Dates: First submitted 2008-03-09; First posted 2008-03-14 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Metastatic Hormone Refractory Prostate Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This study involves the retention of tissue sample from tumor biopsies as well as blood samples.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to look at the genetic changes that RAD001 causes in prostate cancer cells and how those changes relate to patients' response to RAD001 treatment.

DETAILED DESCRIPTION:
This correlative science study will be a minimum risk assessment of tumor and plasma samples collected as part of a Phase II clinical trial of RAD001 in patients with HRPC. Prior to enrollment or at the time of signing consent in the Phase II trial, patients will be approached to participate in the correlative science study. Patients who agree to participate will be assigned a separate study number which will be used to identify their molecular, genetic, genomic and biomarker assessments using the tumor and plasma samples. Clinical outcome results from the accompanying Phase II trial will be used for correlative assessments in this study, however, results from this correlative science study will be kept separate from the assessments and reporting of the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be enrolled in the clinical study entitled: A Single Arm, Phase II Study of RAD001 in Patients with Metastatic, Hormone-Refractory Prostate Cancer at the time of enrollment onto this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult men enrolled in the study entitled: A Single Arm, Phase II Study of RAD001 in Patients with Metastatic, Hormone-Refractory Prostate Cancer.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Functional extent of mTOR inhibition in the phosphorylation status of S6K and CA IX protein in prostate tumors from patients treated with RAD001. | pre-treatment, day 29, and monthly blood samples

SECONDARY OUTCOMES:
To determine by comparative genomic hybridation (CGH) loss of heterozygosity (LOH) patterns of the 10q23 locus (to assess PTEN status) and other sites of chromosomal alterations associated with pathologic response to mTOR inhibition. | pre-treatment, day 19, and monthly blood samples
To identify expression profiles associated with AKT activation and RAD001 treatment effect. | pre-treatment, day 29, and monthly blood samples
To identify candidate plasma markers of glycolysis that reflect tumor AKT activity. | pre-treatment, day 29, and monthly blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J George, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States